CLINICAL TRIAL: NCT00432991
Title: A Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Intramuscular Ephedrine on the Incidence of Perioperative Nausea and Vomiting During Elective Cesarean Section
Brief Title: Study of the Effect of Intramuscular Ephedrine on the Incidence of Nausea and Vomiting During Elective Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0609008727
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Nausea; Vomiting; Cesarean Section
Keywords: Nausea; Vomiting; Cesarean Section
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline Placebo (Placebo Comparator): Drug: Saline Placebo 0.5 mL, IM (in the muscle), one time
  Interventions: Drug: Saline Placebo
- IM Ephedrine (Experimental): Drug: Ephedrine [Synonyms: Ephedra, Ephedrinum] 25 mg, IM (in the muscle), one time
  Interventions: Drug: Ephedrine [Synonyms: Ephedra, Ephedrinum]

INTERVENTIONS:
Drug: Ephedrine [Synonyms: Ephedra, Ephedrinum] — 25 mg, IM (in the muscle), one time
  Arms: IM Ephedrine
Drug: Saline Placebo — 0.5 mL, IM (in the muscle), one time
  Arms: Saline Placebo

SUMMARY:
The purpose of this research study is to investigate if the incidence of nausea and vomiting that subjects experience during and after a Cesarean section can be reduced by giving a shot of the drug ephedrine into the thigh muscle at the time of spinal anesthesia administration.

DETAILED DESCRIPTION:
This research project is designed to study the medication ephedrine, when it is given as a routine part of the anesthesia for elective Cesarean section. Ephedrine is a medication that is widely used in labor and in vaginal and operative (Cesarean section) deliveries to help maintain a woman's blood pressure within its normal range, especially after spinal and epidural anesthesia has been administered. The purpose of this study is to determine if ephedrine, when given intramuscularly (<IM> as a shot in the muscle), at the time of spinal anesthesia administration, can help to decrease the incidence of nausea and vomiting subjects experience during and after a Cesarean section. This study will compare women who receive ephedrine to a similar group of women who receive a normal saline placebo. In addition to looking at the difference in the incidence of nausea and vomiting perioperatively, this study will also evaluate if the administration of IM ephedrine helps the baby to receive more blood from the placenta after anesthesia has been administered to the mother. This will be evaluated by performing a simple blood test, drawn from the umbilical cord, after the baby is born.

ELIGIBILITY:
Inclusion Criteria:

* Must be pregnant with a single baby
* Must be at term in their pregnancy (estimated gestational age of at least 38 weeks)
* Must be scheduled for an elective Cesarean section
* Must be between 60-70" tall
* Must be free of severe systemic disease (ASA class I or II)

Exclusion Criteria:

* Contraindication to spinal anesthesia
* Any allergy to any of the medications included in the study
* History of pregnancy-induced hypertension or preeclampsia
* History of preexisting hypertension
* Diabetes mellitus
* Hyperemesis gravidum
* Previous perioperative nausea and vomiting
* History of motion sickness
* Women carrying a fetus with a known abnormality will also be excluded from the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2007-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Abramovitz, MD, Principal Investigator — Anesthesiology; Weill Medical College of Cornell - New York Presbyterian Hospital
Locations (1):
- New York-Presbyterian Hospital; Weill Medical College of Cornell, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866

RESULTS

PARTICIPANT FLOW:
Groups:
- IM Ephedrine: IM Ephedrine
  Ephedrine [Synonyms: Ephedra, Ephedrinum]: 25 mg, IM (in the muscle), one time
Period: Overall Study
Arm/Group | Saline Placebo | IM Ephedrine
Started | 22 | 31
Completed | 15 | 19
Not Completed | 7 | 12
Not completed — Protocol Violation | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Placebo | IM Ephedrine | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (4.64) | 33.4 (4.4) | 33.7 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pre-Induction Nausea Score
Description: Subject's self-rated nausea level on a scale of 0-3 immediately prior to induction of spinal anesthesia, where 0=no nausea, 1=mild nausea, 2=moderate nausea, and 3=severe nausea
Time Frame: immediately pre-induction
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline Placebo | IM Ephedrine
Number analyzed (Participants) | 15 | 19
units on a scale | 0.067 (0.26) | 0 (0)

2. Primary Outcome: Subject's Self-rated Intra-operative Nausea Level on a Scale of 0-3, Where 0=no Nausea, 1=Mild Nausea, 2=Moderate Nausea, and 3=Severe Nausea.
Description: Subjects were asked to rate their nausea level on a scale of 0-3, where 0=no nausea, 1=mild nausea, 2=moderate nausea, and 3=severe nausea, five times during their procedure: 1) Immediately prior to skin incision, 2) immediately following delivery of the baby, 3) following reinternalization of the uterus, 4) following closure of the fascia, 5) following closure of the skin.
  The numbers given by the subject were then averaged to determine the average level of nausea intra-operatively for each subject.
Time Frame: intra-operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline Placebo | IM Ephedrine
Number analyzed (Participants) | 15 | 19
units on a scale | 0.16 (0.32) | 0.28 (0.34)

3. Primary Outcome: Post-Operation Nausea Score
Description: Subjects were asked to rate their nausea level on a scale of 0-3, where 0=no nausea, 1=mild nausea, 2=moderate nausea, and 3=severe nausea two times after the conclusion of their surgery: 1) upon arrival in the PACU, and 2) immediately prior to discharge from the PACU.
  The numbers given by the subject were then averaged to determine the average level of nausea post-operative for each subject.
Time Frame: post-operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline Placebo | IM Ephedrine
Number analyzed (Participants) | 15 | 19
units on a scale | 0.067 (0.26) | 0.53 (0.77)

ADVERSE EVENTS:
Arm/Group | Saline Placebo | IM Ephedrine
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/31
Other Adverse Events (participants affected / at risk) | 2/22 | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Placebo (N=22) | IM Ephedrine (N=31)
Lightheadedness (General disorders) | 1 (1) | 0 (0)
Pruritis (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes